CLINICAL TRIAL: NCT06254495
Title: A Phase 1, Open-label Study to Evaluate PF-08046044/SGN-35C in Adults With Advanced Malignancies.
Brief Title: A Safety Study of PF-08046044/SGN-35C in Adults With Advanced Cancers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SGN35C-001; C5801001 (Other: Alias Study Number); 2023-505813-26-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Hodgkin Disease; Lymphoma, T-Cell, Peripheral; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Anaplastic
Keywords: cHL; PTCL; sALCL; DLBCL; Seattle Genetics; ADC; Anti Drug Conjugate
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, T-Cell, Peripheral; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Anaplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-08046044/SGN-35C (Experimental): PF-08046044/SGN-35C Monotherapy
  Interventions: Drug: PF-08046044/SGN-35C

INTERVENTIONS:
Drug: PF-08046044/SGN-35C — Given into the vein (IV; intravenously)

SUMMARY:
This clinical trial is studying lymphoma. Lymphoma is a cancer that starts in the blood cells that fight infection. There are several types of lymphoma. This study will enroll people who have classical Hodgkin lymphoma (cHL), peripheral T cell lymphoma (PTCL), or diffuse large B cell lymphoma (DLBCL).

This clinical trial uses a drug called PF-08046044/SGN-35C . The study drug is in testing and has not been approved for sale. This is the first time SGN -35C will be used in people.

This study will test the safety of SGN-35C in participants with lymphoma. It will also study the side effects of this drug. A side effect is anything a drug does to the body besides treating the disease.

This study will have three parts. Parts A and B of the study will find out the best dose and dosing schedule for SGN-35C. Part C will use the dose found in parts A and B to find out how safe SGN-35C is and if it works to treat select lymphomas.

ELIGIBILITY:
Inclusion Criteria:

* Tumor type
* For dose escalation and back fill and dose optimization (Parts A and B):

  * Participants with a histologically confirmed lymphoid neoplasm who in the judgement of the investigator have no appropriate standard therapy available at the time of enrollment and are a candidate for PF-08046044/SGN- 35C treatment. Eligible subtypes and treatment status are as follows:

    * Participants with relapsed/refractory (R/R) cHL: should have received at least 3 prior systemic therapies including autologous stem cell transplant [ASCT] (ASCT and the associated high-dose chemotherapy prior to ASCT are considered to be 1 prior line, along with post-transplant consolidation if progression has not occurred between transplant and start of consolidation) or an anti-PD-1 agent (or refused/were ineligible); or 2 prior systemic therapies if, according to the investigator, no other appropriate standard treatment is available.
    * Participants with R/R PTCL (excluding systematic anaplastic large cell lymphoma [sALCL]): should have received at least 2 prior systemic therapies, or 1 prior systemic therapy if, according to the investigator, no other appropriate standard treatment is available.
    * Participants with R/R sALCL: should have received at least 2 prior systemic therapies, including 1 brentuximab vedotin-containing regimen, or 1 prior line of systemic therapy including brentuximab vedotin, cyclophosphamide, doxorubicin, and prednisone.
    * Participants with R/R DLBCL: should have received at least 2 prior systemic therapies, including ASCT and chimeric antigen receptor (CAR) T-cell therapy, or were ineligible, or refused.
  * Participants with PTCL and DLBCL must have a detectable cluster of differentiation 30 (CD30) expression level (≥1%) in tumor tissue from the most recent biopsy obtained at or after relapse by local testing.
* For dose expansion (Part C):

  * Participants are eligible irrespective of CD30 expression on tumor tissue; however, participants must provide tumor tissue for evaluation of CD30 expression from the most recent biopsy obtained at or after relapse.
  * Participants with cHL, PTCL, sALCL, and DLBCL: Eligible subtypes are the same as defined in Parts A and B
  * If activated, the biology cohort may enroll the populations included in Parts A, B, and C.
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of ≤1
* Fluorodeoxyglucose positron emission tomography (FDG-PET) avid and bidimensional measurable disease as documented by radiographic technique (spiral computed tomography [CT] preferred)

Exclusion Criteria:

* Previous exposure to any antibody-drug conjugates (ADCs) with camptothecin-based payload.
* History of another malignancy within 3 years before the first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy. Exceptions are malignancies with a negligible risk of metastasis or death
* Active central nervous system (CNS) disease related to the underlying malignancy. Participants with a history of CNS disease related to the underlying malignancy are allowed if prior CNS disease has been treated and the participant is clinically stable (defined as not currently receiving steroid treatment for symptoms related to cerebral/meningeal disease and with no ongoing related AE).
* Received previous ASCT infusion <12 weeks prior to the first dose of SGN-35C.
* Previous allogeneic stem cell transplant (SCT) if they meet any of the following criteria:

  * <100 days from allogeneic SCT. Participants ≥100 days from allogeneic SCT who are stable without immunosuppressive therapy for at least 12 weeks are permitted.
  * Active acute or chronic graft-versus-host disease (GVHD) or receiving immunosuppressive therapy as treatment for or prophylaxis against GVHD.
* History of clinically significant GI bleeding, intestinal obstruction, or GI perforation within 6 months of initiation of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2024-05-28 (Actual); Primary Completion 2028-04-18 (Estimated); Study Completion 2029-04-18 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Through 30-37 days after last study treatment, approximately 1 year
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention
Number of participants with laboratory abnormalities | Through 30-37 days after last study treatment, approximately 1 year
Number of participants with dose modifications due to AEs | Up to approximately 1 year
Number of participants with dose-limiting toxicities (DLTs) | Up to 21 days
Number of participants with DLTs by dose level | Up to 21 days

SECONDARY OUTCOMES:
Number of participants with antidrug antibodies (ADA) | Through 30-37 days after last study treatment, approximately 1 year
  To be summarized using descriptive statistics
Area under the concentration time curve (AUC) | Through 30-37 days after last study treatment, approximately 1 year
  To be summarized using descriptive statistics
Maximum concentration (Cmax) | Through 30-37 days after last study treatment, approximately 1 year
  To be summarized using descriptive statistics
Time at which the maximum concentration occurs (Tmax) | Through 30-37 days after last study treatment, approximately 1 year
  To be summarized using descriptive statistics
Apparent terminal half-life (t1/2) | Through 30-37 days after last study treatment, approximately 1 year
  To be summarized using descriptive statistics
Trough concentration (Ctrough) | Through 30-37 days after last study treatment, approximately 1 year
  To be summarized using descriptive statistics
Objective response rate (ORR) as assessed by the investigator | Up to approximately 1 year
  A participant is determined to have an objective response if, based on Lugano criteria (Cheson 2014), they achieve a complete response (CR) or partial response (PR) as assessed by the investigator. The ORR is defined as the percentage of participants with an objective response.
CR rate as assessed by the investigator | Up to approximately 1 year
  CR rate is defined as the proportion of participants with CR.
Duration of response (DOR) | Up to approximately 1 year
  DOR is defined as the time from the start of the first documentation of objective tumor response (CR or PR) to the first documentation of tumor progression per Lugano criteria (Cheson 2014) as assessed by the investigator or to death due to any cause, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (33):
- United States (27):
  - City of Hope (City of Hope National Medical Center, City Of Hope Medical Center), Duarte, California
  - IP Address: City of Hope Investigational Drug Services(IDS), Duarte, California
  - University of California, San Francisco Medical Center, San Francisco, California
  - Sylvester Comprehensive Cancer Center- The Lennar Foundation Medical Center, Coral Gables, Florida
  - University of Miami Hospital and Clinics - Deerfield Beach, Deerfield Beach, Florida
  - Sylvester Comprehensive Cancer Center - Hollywood, Hollywood, Florida
  - University Of Miami Hospital and Clinics/Sylvester Comprehensive Cancer Center, Miami, Florida
  - University Of Miami Hospitals And Clinics, Miami, Florida
  - Sylvester Comprehensive Cancer Center - Kendall, Miami, Florida
  - The University of Kansas Cancer Center, Investigational Drug Services, Fairway, Kansas
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - The University of Kansas Hospital Cambridge North Tower A, Kansas City, Kansas
  - The University of Kansas Hospital, Kansas City, Kansas
  - The University of Kansas Medical Center Medical Office Building, Kansas City, Kansas
  - The University of Kansas Cancer Center - Overland Park, Overland Park, Kansas
  - The University of Kansas Cancer Center - Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Cancer Center, Westwood, Kansas
  - The University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Nebraska Medicine - Bellevue Medical Center, Bellevue, Nebraska
  - Nebraska Medical Center, Omaha, Nebraska
  - Nebraska Medicine - Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - Fred Hutchinson Cancer Research Center | Seattle, WA, Seattle, Washington
  - University of Washington, Seattle, Washington
- Rigshospitalet University Hospital of Copenhagen, Copenhagen Ø, Denmark
- Institut Gustave Roussy, Villejuif, France
- Centro Ricerche Cliniche di Verona s.r.l., Verona, Italy
- Hospital Universitari Vall d'Hebron, Barcelona, Spain
- United Kingdom (2):
  - The Royal Marsden NHS Foundation Trust (RM), London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SGN35C-001